CLINICAL TRIAL: NCT07396532
Title: Nurse-Led Audio-Recorded Reorientation to Reduce Delirium in Elderly Hip Fractures: A Pilot Randomized Control Trial
Brief Title: Audio-Recorded Messages Delivered Via iPad to Prevent Delirium in Hip Fracture Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-0733; CIRB-2025-0733 (Registry Identifier: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2025-12-03; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Delirium - Postoperative; Delirium and Post-operative Cognitive Dysfunction (POCD); Delirium, Postoperative
Keywords: delirium; nurse-led; reality reorientation; AI
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: Group 1 (intervention group): Audio reorientation intervention + usual care Group 2 (control group): Usual care only Both groups studied simultaneously with the same time period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-Recorded Reorientation Intervention (Experimental): Participants in this arm receive personalized audio-recorded reorientation messages delivered three times daily during the first three post-operative days. Each message lasts approximately 2 minutes and contains personalized information including the current location, date and time, and encouraging messages. Messages are delivered via iPad and headphones by nursing staff during routine care. Audio messages are available in English, Mandarin, Malay, and Tamil to accommodate patient language preferences. Participants also receive all standard post-operative care and treatments.
  Interventions: Behavioral: Audio-Recorded Reorientation Intervention
- Standard Care Control (No Intervention): Participants in this arm receive standard hip fracture care according to the hospital's established hip fracture pathway. Standard care includes early mobilization with sitting out of bed three times daily, allied health professional involvement (physiotherapist, occupational therapist, and dietitian), and routine orientation assessment.
  Participants found to be disoriented are screened for delirium using the validated 4AT assessment tool administered by nursing staff. Those identified as at-risk or experiencing delirium receive a comprehensive delirium care bundle including environmental modifications, medication review, and enhanced monitoring. Standard reorientation interventions include whiteboard orientation displays and purple wrist tags for participants at risk of cognitive impairment to ensure enhanced monitoring and fall prevention.
  No study-specific interventions are provided to this group beyond routine hospital care protocols.

INTERVENTIONS:
Behavioral: Audio-Recorded Reorientation Intervention — Participants in this arm receive personalized audio-recorded reorientation messages delivered three times daily during the first three post-operative days. Each message lasts approximately 2 minutes and contains personalized information including the current location, date and time, and encouraging messages. Messages are delivered via iPad and headphones by nursing staff during routine care. Audio messages are available in English, Mandarin, Malay, and Tamil to accommodate patient language preferences. Participants also receive all standard post-operative care and treatments.
  Arms: Audio-Recorded Reorientation Intervention

SUMMARY:
The goal of this pilot clinical trial is to learn if personalized audio-recorded reorientation messages can be successfully implemented in general hospital wards for elderly patients after hip fracture surgery. It will also explore whether this intervention might help prevent confusion (delirium) after surgery. The main questions it aims to answer are:

* Can the intervention be successfully delivered by nursing staff in a busy orthopedic ward?
* How many eligible patients can be recruited and retained in the study?
* Do patients tolerate listening to the personalized audio messages without problems?
* Does listening to personalized audio messages show any early signs of reducing confusion after surgery?

Researchers will compare patients who receive personalized audio messages to those who receive usual care to see if the intervention is feasible to implement and whether it shows promise for preventing delirium.

Participants will:

* Listen to 2-minute personalized audio-recorded reorientation messages played through an iPad and headphones three times daily for the first 3 days after surgery
* Have their orientation and mental status checked daily for three times by nursing staff
* Continue with all their regular medical care and treatments
* Be monitored until discharge from the study wards.

DETAILED DESCRIPTION:
Background and Rationale:

Hip fracture surgery is common among elderly patients, but recovery can be complicated by post-operative delirium (confusion), which affects up to 50% of patients and can lead to longer hospital stays, increased complications, and delayed rehabilitation. Non-pharmacological interventions, particularly reorientation strategies, have shown promise in preventing delirium, but implementation in busy hospital wards remains challenging.

Study Design and Innovation:

This pilot randomized controlled trial tests an innovative approach using personalized audio-recorded reorientation messages delivered via 'Shortcut' Application on the iPad technology. The messages are available in multiple languages (English, Mandarin, Malay, Tamil) to accommodate the diverse patient population, but the content is standardized across all participants. This technology-supported approach enables nurses to provide systematic reorientation interventions as part of their routine care.

Intervention Details:

The audio messages are approximately 2 minutes long and include: reorientation information (patient's location, real-time update of date and time, reason for admission), explanation of their recovery process, encouragement for therapy participation, pain management guidance, and reassuring messages on who are taking care of them in the hospital. Messages are played through noise-canceling headphones to ensure clarity and minimize ward noise interference.

Implementation Approach:

Nursing staff receive brief training on the iPad system and the workflow process. The intervention is designed to be sustainable within existing workflow patterns without adding significant burden to clinical staff. Visual reminders of workflow process were also readily available in nursing stations to remind the nurses. Study team also do their rounds to ensure availability of equipment and to clarify doubts from nursing staff.

Target Population:

Elderly patients (≥60 years) admitted to orthopedic wards following hip fracture surgery who are at risk for developing post-operative delirium based on established risk factors.

Feasibility Focus:

As a pilot study, this research prioritizes understanding implementation challenges, staff acceptance, patient tolerance, and recruitment feasibility to inform the design of a future definitive trial examining delirium prevention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60 years and above
* Undergoing hip fracture repair surgery
* No history of cognitive impairment as assessed by Abbreviated Mental Test (AMT)
* Able to understand to any of the basic languages of Singapore (English, Malay, Mandarin, Tamil)

Exclusion Criteria:

* Patients not admitted directly to orthopaedic (study) wards post-operation (such as those requiring post-operative high-dependency unit care)
* Patients managed conservatively without surgical intervention.
* Patients admitted for periprosthetic hip fracture repairs
* Patients who are deaf and mute

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Protocol Adherence Rate | Postoperative day 1 to postoperative day 3
  Percentage of planned audio-recorded reorientation sessions successfully delivered by the nurses across the first 3-day intervention period. Target adherence rate ≥95% to demonstrate intervention feasibility.
Recruitment Feasibility | From enrollment to end of study participation (up to 2 weeks)
  Recruitment feasibility measured by screening-to-enrollment rate, calculated as: (1) percentage of screened patients meeting eligibility criteria, and (2) percentage of eligible patients providing informed consent. These rates will be tracked throughout the study period to assess the feasibility of recruiting the target population for a future definitive trial. Target enrollment rate of ≥80% of eligible patients will indicate feasibility.
Study Retention Rate | From enrollment to end of study participation (up to 2 weeks)
  Percentage of enrolled participants who completed the study protocol without withdrawal, calculated as number completing study divided by total enrolled. Target retention rate ≥90% to demonstrate intervention feasibility.
Intervention Tolerance Rate | Postoperative Day 1 to Postoperative Day 3
  Completion of each audio-recorded reorientation session without early discontinuation or adverse reactions, assessed during each of the 9 planned sessions per participant. Target adherence rate ≥95% to demonstrate intervention feasibility.

SECONDARY OUTCOMES:
Number of participants with delirium as assessed by 4AT (4 'A's Test) screening tool | From postoperative day 1 to end of study participation (up to 2 weeks)
  Delirium will be assessed using the 4AT (4 'A's Test), a validated 4-item screening instrument that evaluates alertness, attention (months backwards), acute change or fluctuating course, and AMT4 (age, date of birth, place, current year). The 4AT score ranges from 0-12, with scores ≥4 indicating possible delirium and scores ≥1 suggesting cognitive impairment. Delirium incidence will be reported as the number and percentage of participants who score ≥4 on the 4AT during their study participation period.
Length of stay in study ward measured in days | From admission to pilot ward until discharge/transfer from pilot ward (up to 2 weeks)
  Length of stay will be measured as the total number of days from admission to the pilot ward until discharge from the pilot ward (either to home, transfer to another ward, or transfer to community hospital). This measure captures only the time spent specifically in the study/pilot ward and does not include any subsequent stays in other wards or facilities. Length of stay will be calculated in whole days and reported as mean, median, and range.
Number of participants actively participating in prescribed physiotherapy and occupational therapy sessions | From postoperative day 1 to postoperative day 3
  Allied health participation will be measured as the number and percentage of participants who actively engage in their prescribed physiotherapy (PT) and occupational therapy (OT) sessions during their stay in the pilot ward. Participation will be defined as attending and actively engaging in therapy sessions as documented by the treating therapists. Since all hip fracture patients receive standard PT/OT orders, this outcome measures engagement rather than referral rates. Data will be collected through therapy documentation review.
Cumulative analgesic consumption | From postoperative day 1 to postoperative day 3
  Analgesic consumption will be measured as the total cumulative dose of commonly prescribed analgesics (morphine, paracetamol, and oxycodone) consumed by participants during post-operative days 1 to 3. All doses will be recorded in their respective units (morphine in mg, paracetamol in mg, oxycodone in mg) from medication administration records. This outcome assesses whether improved orientation and medication compliance messaging through the audio-recorded intervention affects analgesic usage patterns. Data will include both scheduled and PRN (as needed) doses administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the pilot nature of this feasibility study with a small sample size. Aggregate results and study findings will be made available through peer-reviewed publications and conference presentations. The study protocol and statistical analysis plan will be made publicly available.

REFERENCES:
- [Background] Munro CL, Cairns P, Ji M, Calero K, Anderson WM, Liang Z. Delirium prevention in critically ill adults through an automated reorientation intervention - A pilot randomized controlled trial. Heart Lung. 2017 Jul-Aug;46(4):234-238. doi: 10.1016/j.hrtlng.2017.05.002. Epub 2017 Jun 9. PMID 28606450
- [Background] Kasapoglu ES, Enc N. Role of multicomponent non-pharmacological nursing interventions on delirium prevention: A randomized controlled study. Geriatr Nurs. 2022 Mar-Apr;44:207-214. doi: 10.1016/j.gerinurse.2022.02.015. Epub 2022 Feb 26. PMID 35227973